CLINICAL TRIAL: NCT04985786
Title: Pathological Risk: Dynamics of Risk Perception and Risk Behavior in Alcohol Use Disorder and Schizophrenia
Brief Title: Dynamics of Risk Perception and Risk Behavior in Alcohol Use Disorder and Schizophrenia
Acronym: PathRisk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Konstanz (Other)
Collaborators: Centre for Psychiatry Reichenau, Germany (Unknown)
Responsible Party: Principal Investigator, Michael Odenwald, Chief Psychologist Research Ward, University of Konstanz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OD 113/3-1
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Alcohol Use Disorder (AUD); Schizophrenia and Related Disorders
MeSH Terms: conditions — Alcoholism; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AUD Intervention (Experimental): Risk behavior specific intervention, targeting alcohol drinking
  Interventions: Behavioral: Cognitive Behavioral Therapy for reducing risk behaviors
- AUD Control (Active Comparator): Non-risk behavior specific intervention, targeting cognitive exercises
  Interventions: Behavioral: Cognitive Behavioral Therapy for increasing non-risk behaviors
- AUD & SZ Intervention (Experimental): Risk behavior specific intervention, targeting alcohol drinking
  Interventions: Behavioral: Cognitive Behavioral Therapy for reducing risk behaviors
- AUD & SZ Control (Active Comparator): Non-risk behavior specific intervention, targeting cognitive exercises
  Interventions: Behavioral: Cognitive Behavioral Therapy for increasing non-risk behaviors
- SZ Intervention (Experimental): Risk behavior specific intervention, targeting medication non-adherence
  Interventions: Behavioral: Cognitive Behavioral Therapy for reducing risk behaviors
- SZ Control (Active Comparator): Non-risk behavior specific intervention, targeting cognitive exercises
  Interventions: Behavioral: Cognitive Behavioral Therapy for increasing non-risk behaviors
- HC Control (No Intervention): Healthy control subjects will participate in fMRI assessments only

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for reducing risk behaviors — Cognitive Behavioral Therapy to reduce risk behaviors and increase risk perception that combines a standardised face-to-face group therapy before discharge from in-patient treatment and a standardised ecological momentary intervention delivered by mobile phones during the four weeks after discharge. For SZ the target risk behavior is medication non-adherence and for AUD and AUD & SZ it is alcohol use.
  Arms: AUD & SZ Intervention; AUD Intervention; SZ Intervention
Behavioral: Cognitive Behavioral Therapy for increasing non-risk behaviors — Cognitive Behavioral Therapy to increase non-risk behaviors that combines a standardised face-to-face group therapy before discharge from in-patient treatment and a standardised ecological momentary intervention delivered by mobile phones during the four weeks after discharge. In this control intervention for patient groups the target behavior is cognitive exercises.
  Arms: AUD & SZ Control; AUD Control; SZ Control

SUMMARY:
The hyper- or hypo-attribution of risks is deeply related to the core pathological mechanisms of mental disorders and at the same time engaging in risky behaviors influences their course and outcomes. The investigators study risk perception, risk behaviors and underlying brain mechanisms in a longitudinal design in three groups of psychiatric patients who participate in a psychological intervention that is aimed to reduce risk behavior and increase risk perception.

Patients with schizophrenia (SZ), alcohol use disorder (AUD) and both disorders (SZ + AUD) are recruited during psychiatric in-patient treatment and participate in a combined face-to-face and mobile intervention that starts before release and ends four weeks after discharge. The standardized 4-session face-to-face group intervention that is based on motivational interviewing (Miller & Rollnick, 2013) and relapse prevention (Marlatt & Donovan, 2005) and addresses the reduction of disorder-specific risk behaviors, i.e. alcohol use for AUD and SZ+AUD and medication non-adherence for SZ. After discharge, a 4-week ecological momentary intervention (EMI) supports participants to maintain abstinence from risk behaviors and to strengthen coping in high-risk situations relying on mental contrasting and implementation intentions (Oettingen & Gollwitzer, 2011). Participants will be assessed in fMRI and behavioral measurements and by self-report pre and post interventional phase, furthermore they participate in an ecological momentary assessment during the post-discharge phase which assesses risk behaviors, high-risk situations and risk perception in real life contexts.

ELIGIBILITY:
Inclusion Criteria:

* for patient groups: fulfilling the diagnostic criteria for AUD or SZ or both

Exclusion Criteria:

for patient groups and healthy control group:

* no sufficient command of German language
* neurological disorder for patient groups:
* acute psychotic episode
* acute suicidality or not distanced from self-harming behaviors
* other substance use disorder (exception: nicotine and caffeine use disorders) for healthy control group:
* absence of any psychiatric diagnosis (exception: nicotine and caffeine use disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of Nucleus Accumbens activation and connectivity during risky decision making | 6 weeks
  Change of fMRI signal (BOLD) in Balloon Analogue Risk Task
Engagement in risk behaviors | 4 weeks
  Alcohol drinking (for AUD and AUD+SZ) and medication non-adherence (for SZ) as recorded by ecological momentary assessment (EMA)

SECONDARY OUTCOMES:
Risk reappraisal | 4 weeks
  Change of risk perception after critical event depending on the outcome of the critical event (engaging is risk behavior or not) as defined by Klepper et al. (2017)
Activation of amygdala, STS, mPFC and insula during risk evaluation | 6 weeks
  fMRI signal (BOLD) in a trustworthiness task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Konstanz, Research Ward, Konstanz, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request ensuring the data protection laws are fulfilled
Time Frame: 6 months after publication
Access Criteria: will be defined according to legal requirements

REFERENCES:
- [Background] Klepper S, Odenwald M, Rosner S, Senn S, Menning H, Pereyra-Kroll D, Rockstroh B. Experience-Induced Change of Alcohol-Related Risk Perception in Patients with Alcohol Use Disorders. Front Psychol. 2017 Nov 13;8:1967. doi: 10.3389/fpsyg.2017.01967. eCollection 2017. PMID 29180975
- [Background] Gollwitzer P, Oettingen G (2011). Planning promotes goal striving. In: KD Vohs, RF Baumeister (Eds.), Handbook of Self-Regulation: Research, Theory, and Applications (2nd edition, chapter 9, pp. 162 - 184). The Guilford Press.
- [Background] Marlatt GA, Donovan, DM. Relapse Prevention. 2nd edition. The Guilford Press.
- [Background] Miller R, Rollnick S (2013) Motivational Interviewing. 3rd edition. The Guilford Press.